CLINICAL TRIAL: NCT05085600
Title: Effects of a Single Manual Therapy-Exercise Versus Exercise Session in Patients With Chronic Neck Pain and Upper Cervical Spine Dysfunction. Randomized Controlled Trial
Brief Title: Effects of a Single Manual Therapy-Exercise Versus Exercise Session in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER-2021-A2
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Neck Pain
Keywords: spine; manual therapy; exercise; chronic neck pain
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): 20-minute session, composed of 2 blocks of 10 repetitions, holding each exercise for 10 seconds, a 40-second rest between each repetition and 2 minutes between blocks.
  Interventions: Other: Exercise
- Exercise + Manual Therapy Group (Experimental): 20-minute session. In the first 5 minutes, muscle techniques will be performed to prepare the tissue of the upper cervical spine before applying joint techniques. In the next 15 minutes, manipulation and / or mobilization techniques of the upper cervical spine, including the C2-3 segment, will be combined with cervical exercise
  Interventions: Other: Manual Therapy + Exercise

INTERVENTIONS:
Other: Exercise — Patients will begin performing the cervical stabilization exercise, and will taught to perform the contraction of deep neck flexor muscle activity with the help of the Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) in supine.
  In addition, progress will continued in the exercise of the contraction of deep neck flexor muscles in other positions.
  The progression of the exercises will be adapted to each patient, depending on their evolution. Firstly, exercises will undertaken in the supine and standing positions; once these positions will mastered, the exercises progressed to asymmetric positions with cervical bending and/or rotation toward each patient's most symptomatic side.
  Arms: Exercise Group
Other: Manual Therapy + Exercise — 20-minute session. In the first 5 minutes, muscle techniques will be performed to prepare the tissue of the upper cervical spine before applying joint techniques. In the next 15 minutes, manipulation and / or mobilization techniques of the upper cervical spine, including the C2-3 segment, will be combined with cervical exercise
  Arms: Exercise + Manual Therapy Group

SUMMARY:
Chronic neck pain is described as pain located between the occiput and the third thoracic vertebra that persists for more than 3 months. Chronic neck pain is one of the biggest musculoskeletal health problem in industrialized countries, representing 14.6% of all such problems today. 50% of the adult population will experience cervical pain at some point during the year.

The objective of this study is to compare the effectiveness of a single exercise session with manual therapy techniques of the upper cervical spine against a single exercise session in patients with chronic neck pain and upper cervical spine dysfunction.

The treatment will be applied by 1 therapist with orthopedic manual therapist (MT)-specialist training and more than 10 years of MT experience.

The primary outcome measurements will be cervical mobility and cervical pressure pain threshold. Intensity of pain will be also used as secondary outcome measure. These measurements shall be taken before and immediately after the relevant intervention.

Exercise Group After the baseline assessments, patients will performed the cervical stabilization exercise, and will taught to perform the contraction of deep neck flexor muscle activity with the help of the Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) in supine.

In addition, progress will continued in the exercise of the contraction of deep neck flexor muscles in other positions.

The progression of the exercises will be adapted to each patient, depending on their evolution. Firstly, exercises will undertaken in the supine and standing positions; once these positions will be mastered, the exercises progressed to asymmetric positions with cervical bending and/or rotation toward each patient's most symptomatic side. Also, no pain will be allowed in the positions. Exercises were always carried out without pain, because pain can be an inhibitor of muscle contraction.

The Exercise (E) group will carried out one 20-minute session, composed of 2 blocks of 10 repetitions, holding each exercise for 10 seconds, a 40-second rest between each repetition and 2 minutes between blocks.

Manual Therapy + Exercise Group The MT + E group will carried out 20-minute sessions led by an experienced physical therapist. In the first 5 minutes, muscle techniques will be performed to prepare the tissue of the upper cervical spine before applying joint techniques. In the next 15 minutes, manipulation (high velocity low amplitude) and / or mobilization techniques of the upper cervical spine, including the C2-3 segment, will be combined with cervical exercise. The MT techniques were applied depending on the clinical findings in each patient.

DETAILED DESCRIPTION:
Chronic neck pain is described as pain located between the occiput and the third thoracic vertebra that persists for more than 3 months. Chronic neck pain is one of the biggest musculoskeletal health problem in industrialized countries, representing 14.6% of all such problems today. 50% of the adult population will experience cervical pain at some point during the year.

The objective of this study is to compare the effectiveness of a single exercise session with manual therapy techniques of the upper cervical spine against a single exercise session in patients with chronic neck pain and upper cervical spine dysfunction.

The treatment will be applied by 1 therapist with orthopedic manual therapist (MT)-specialist training and more than 10 years of MT experience.

The primary outcome measurements will be cervical mobility and cervical pressure pain threshold. Intensity of pain will be also used as secondary outcome measure. These measurements shall be taken before and immediately after the relevant intervention.

Exercise Group After the baseline assessments, patients will performed the cervical stabilization exercise, and will taught to perform the contraction of deep neck flexor muscle activity with the help of the Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) in supine.

In addition, progress will continued in the exercise of the contraction of deep neck flexor muscles in other positions.

The progression of the exercises will be adapted to each patient, depending on their evolution. Firstly, exercises will undertaken in the supine and standing positions; once these positions will be mastered, the exercises progressed to asymmetric positions with cervical bending and/or rotation toward each patient's most symptomatic side. Also, no pain will be allowed in the positions. Exercises were always carried out without pain, because pain can be an inhibitor of muscle contraction.

The Exercise (E) group will carried out one 20-minute session, composed of 2 blocks of 10 repetitions, holding each exercise for 10 seconds, a 40-second rest between each repetition and 2 minutes between blocks.

Manual Therapy + Exercise Group The MT + E group will carried out 20-minute sessions led by an experienced physical therapist. In the first 5 minutes, muscle techniques will be performed to prepare the tissue of the upper cervical spine before applying joint techniques. In the next 15 minutes, manipulation (high velocity low amplitude) and / or mobilization techniques of the upper cervical spine, including the C2-3 segment, will be combined with cervical exercise. The MT techniques were applied depending on the clinical findings in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with chronic neck pain
* More than 18 years old
* Loss of mobility in one or more upper cervical spine segments found through manual assessment according to Zito et al. (2006) and Kaltenborn (2012).
* A positive result in the Flexion rotation-test in the upper cervical spine (less than 32º or a difference of 10º or more between the two rotations.
* Not being able to exceed 24 mmHg in the cranio-cervical flexion test.
* Signing the informed consent.

Exclusion Criteria:

* Contraindication to manual therapy or exercise (pathological changes due to neoplasm, inflammation infections, osteopenia, congenital collagenous compromise syndromes "Down´s, Ehlers-Danlos, Grisel, Morquio"
* Marked degeneration of the cervical spine that may affect cervical spine ligament integrity.
* History of trauma to cervical vessels.
* Anticoagulant therapy or blood clotting disorders or to have participated in any program of exercises or manual therapy treatments designed to improve the performance of the cervical region in the previous 3 months.
* Post-traumatic neck pain or red flags according to Rushton et al.
* Inability to maintain the supine position, use of pacemakers, an inability to perform the flexion rotation-test
* Language difficulties that hinder understanding of informed consent or completion of the questionnaires necessary for this study.
* Subjects with litigation or lawsuits pending

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Active range of motion mobility in the inferior cervical region (º) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Mobility in the inferior cervical region will be evaluated in a sitting position with the back vertical and resting on the backrest of the chair with a CROM device (floating compass; Plastimo Airguide, Inc, Buffalo Groove,IL). Flexion, extension, right and left side-bending and right and left rotation will be measured. Three measurements will be made for each movement, and the result will be the mean of the three measurements.
Active range of motion mobility in the upper cervical region (º) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Flexion rotation-test will be used to measure the upper rotation, predominantly at C1-2. To perform this test, the subjects position themselves in the supine position and the evaluator passively will take the patients cervical spine to its maximum flexion and then will rotated the head to the right and left side with the occiput resting against the evaluator's abdomen. The movement will stopped at whichever situation occurs first, either the subject presents symptoms, or the evaluator reaches the end of the range of motion and finds a firm end feel. A CROM device will be used too, and three measurements will be performed for each movement, with the result being the mean of the three measurements
Pressure Pain Threshold (Kpa) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Cervical pressure pain threshold (PPT) will be measured using a digital algometer (Somedic AB Farsta, Somedic SenseLab AB, Sweden) with a round surface area of 1 cm2, and pressure will be applied at the rate of 1 kg/cm2/s perpendicular to the skin. With the subject supine, PPT will be assessed over 6 points bilaterally with a 10-second rest between each measurement: first metacarpal joint, upper trapezius muscle, elevator of scapula, C5-6 zygapophyseal joint, C2-3 zygapophyseal joint, and suboccipital muscles. Patients will be instructed to press the button of the digital algometer at the precise moment that pressure sensation changed to pain. The mean of 3 trials will be calculated over each point and used for analysis.

SECONDARY OUTCOMES:
Pain Intensity (Visual analogue scale 0-100 mm) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Intensity of pain in the cervical region will be measured with VAS from 0 to 100 mm in length, with the extremes defined as "no pain" (0) and "the worst pain imaginable" (100) and without any intermediate points.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain